CLINICAL TRIAL: NCT00006393
Title: Genetic Study of the FBN1 Gene and Fibrillin-1 Abnormalities in Choctaw Native Americans and Other Patients With Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Other Study IDs: NCRR-M01RR02558-0104; UT-H-HSC-MS-96-206
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Systemic Sclerosis
Keywords: arthritis & connective tissue diseases; rare disease; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Arthritis; Connective Tissue Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Determine whether defects in fibrillin-1 cellular processing are present in the tsk1 mouse model that carries a known FBN1 gene rearrangement and in a population of Choctaw Native American patients with systemic sclerosis who have a strong genetic predisposition to the disease.

II. Determine the ultrastructural features of fibrillin-1 in these patients. III. Screen the FBN1 gene for mutations beginning at the regions homologous to the tsk1 duplication and latent transforming growth factor binding proteins in these patients and in an unaffected Choctaw control group.

IV. Determine the correlation between fibrillin-1 abnormalities and clinical presentation, autoantibodies, and ethnicity.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients undergo punch skin biopsy obtained from the upper arm or back. Studies of fibrillin-1 synthesis and cellular processing, and FBN1 mutational analysis, linkage analysis, and genetic mapping are performed on the tissue samples. Patients from all major US ethnic groups (Caucasian, Hispanic, African Americans) will be recruited for the study in the next 2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of systemic sclerosis in accordance with the American College of Rheumatology preliminary criteria

Positive for systemic sclerosis antibodies (e.g., anticentromere, antitopo, antifibrillarin, or antiRNA polymerase)

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Filemon Tan, M.D., Study Chair — University of Texas
Locations (1):
- University of Texas- Houston Medical School, Houston, Texas, United States